CLINICAL TRIAL: NCT03809897
Title: An Effectiveness and Safety Study of Varenicline for Smoking Cessation in Hospitalized Patients With Psychiatric Disorders
Brief Title: Varenicline for Smoking Cessation in Hospitalized Patients With Psychiatric Disorders
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Budget not sufficient to cover the study scope proposed and recruitment rates expected to be no sufficient.
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Clínica Galatea (Unknown); Hospital Sant Rafael (Unknown); Hospital de Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRU-VCN-2017
Record Dates: First submitted 2018-11-21; First posted 2019-01-18 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-01

CONDITIONS: Tobacco Use Cessation; Psychiatric Disorders
MeSH Terms: conditions — Tobacco Use Cessation; Mental Disorders | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive varenicline or nicotine patch during 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varenicline (Experimental): Patients randomized to the experimental arm will receive 3 days of 0.5 mg of varenicline, followed by 4 days of 1 mg of varenicline (until day 7). Finally, until week 12, they will receive 2 mg of varenicline. Varenicline is supplied in capsules and taken orally.
  Interventions: Drug: Varenicline
- Nicotine patch (Active Comparator): Patients randomized to nicotine patch will receive 8 weeks of 21 mg patch followed by 2 weeks of 14 mg patch and 2 weeks of 7 mg patch.
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Varenicline — All participants randomized to varenicline will be titrated to the full dose during the first week and continued up to week 12 following standard dosage. This would be independent of time of discharge, so patients will continue the same treatment after discharge up to complete the 12 weeks.
  Other Names: Champix
  Arms: Varenicline
Drug: Nicotine patch — Patients randomized to nicotine patch will receive 8 weeks of 21mg patch followed by 2 weeks of 14 mg patch and 2 weeks of 7 mg patch.
  Other Names: Nicotinell
  Arms: Nicotine patch

SUMMARY:
Varenicline increases smoking abstinence rates compared to bupropion, nicotine patch or placebo in outpatients with psychiatric disorders. The American Psychiatric Association identifies psychiatric hospitalizations as an ideal opportunity to treat tobacco dependence. However, no previous studies have tested whether varenicline may improve smoking cessation rates compared to nicotine patch in hospitalized patients with mental illness. Additionally, varenicline has shown to be safe for mental health stable outpatients, but safety in psychiatric inpatients is unknown.

Multisite open trial controlled study designed to assess varenicline's effectiveness on smoking cessation compared to nicotine patch, in patients who are discharged from a psychiatric unit. Treatment will start during hospitalization and last 12 weeks followed by a non-treatment follow-up phase for 4 weeks. Safety will be assessed by comparing the incidence of adverse events.

Participants will be randomized to receive varenicline or nicotine patch during 12 weeks. All participants will receive smoking cessation counseling.

DETAILED DESCRIPTION:
Varenicline has shown to increase abstinence rates compared to other pharmacological interventions (including nicotine patch) or placebo in outpatients with psychiatric disorders. Safety of varenicline in this population has also been stated as adverse events are similar to other smoking cessation medications.

Taking into account that varenicline has shown to increase abstinence rates in outpatients with psychiatric disorders compared to other smoking cessation medications, and no previous studies have measured the impact of initiating varenicline during psychiatric hospitalization, this study will compare varenicline to nicotine patch initiated during hospitalization on smoking abstinence rates (treatment will last 12 weeks; and there will be additional 4 weeks of non-treatment).

Regarding safety, inpatient wards are probably the best setting to test safety as any adverse effect can be reported immediately and in case of an intervention needed, this can be provided at once.

This study will have three phases: screening phase (1), treatment phase (2a and 2b), and non-treatment phase (3).

1. Screening phase: Psychiatrists and psychologists will be responsible for informing to potential participants about the study, and check eligibility for each patient. Investigators will give informed consent and information sheet to the participant, and all doubts will be resolved appropriately. If subject decides to participate the informed consent will be signed. The screening period will take place during first 72 hours after admission and participants will be randomized before 96 hours after admission.
2. Treatment phase: Treatment will take 12 weeks, therefore varenicline and nicotine patch will be dispensed during hospitalization and after discharge up to complete 12 weeks. All participants randomized to varenicline will be titrated to the full dose during the first week and continued up to week 12 following standard dosage. This would be independent of time of discharge, so patients will continue the same treatment after discharge up to complete the 12 weeks. Patients randomized to nicotine patch will receive 8 weeks of 21mg patch followed by 2 weeks of 14 mg patch and 2 weeks of 7 mg patch.

   1. During hospitalization: All participants will be assessed regarding their psychiatric and drug use history (including smoking) as well as past and current psychiatric disorders diagnosed by their psychiatrist. Adverse events (volunteered, observed, or solicited) will be also evaluated and recorded by their psychiatrist. Serious adverse events will be considered as an untoward medical occurrence at any dose that results in death, or is life-threatening, or requires prolongation of the hospitalization, or results in persistent or significant disability/incapacity, or results in congenital anomaly birth defect (following the same criteria of other studies). In case of serious adverse events (SAEs) at any point of the study, Principal Investigators will report to Pfizer within 24 hours of first awareness of the event. Cigarette Dependence, Tobacco withdrawal, Global Clinical Impression, nicotine use, suicide ideation/behavior, anxiety and depression will be assessed via scales and questionnaires by a trained smoking cessation psychologist. This psychologist will be also in charge of delivering weekly a motivationally tailored smoking cessation group counseling (30-45 minutes) following an adaptation of the manualized curriculum. A nurse will be responsible for measuring the end-expiratory exhaled CO, record body height and weight, vital signs (blood pressure and heart rate) and dispense medication.
   2. After discharge: There will be weekly visits until week 5, and visits at weeks 7, 9 and 12. Post-hospitalization visits will include tobacco use assessment, mental health assessment, adverse-events assessment, smoking cessation counseling and varenicline or nicotine patch delivery up to following visit. A psychiatrist will be responsible for assessing adverse-events and mental health. A psychologist will be responsible for delivering smoking cessation counseling tailored to each participant's needs according to the manualized curriculum and assessing tobacco use, withdrawal, suicide ideation/behavior, Global Clinical Impression, anxiety and depression. Counseling and mental health assessment will be conducted by the same professional whenever possible. A nurse will be responsible for measuring the end-expiratory exhaled CO, record body weight, vital signs (blood pressure and heart rate) and dispense medication. Whenever participant does not attend a study visit, counseling and Nicotine Use Inventory (NUI) will be delivered by telephone.
3. Non-treatment phase: This will include a telephone visit at week 14 and a face-to-face visit at week 16. Telephone visit will be made by the psychologist and it will include tobacco use assessment and smoking cessation counseling. A psychiatrist will be responsible for assessing adverse-events and mental health at week 16 visit and a psychologist will assess tobacco use, withdrawal, suicide ideation/behavior, Global Clinical Impression, anxiety and depression, and deliver smoking cessation counseling. Counseling and mental health assessment will be conducted by the same professional whenever possible. Also at this point,an End-of-study questionnaire will be completed. A nurse will be responsible for measuring the end-expiratory exhaled CO, record body weight and vital signs (blood pressure and heart rate). Whenever participant does not attend a study visit, NUI will be delivered by telephone. In case of early termination at any point of the study, an End-of-study questionnaire will be also completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years old, inclusive.
2. Good understanding of protocol to informed consent.
3. Hospitalized for a mental health condition at one of the three acute psychiatric facilities who participate in this study.
4. Having at least a psychiatric disorder according to DSM-5.
5. Living in Barcelona city or in the metropolitan area.
6. Not being at high risk of self-injury or suicidal behavior, in the opinion of the Investigator.
7. Smoking an average of at least 10 cigarettes per day during the year before hospital admission.
8. Females who are not childbearing potential (surgical sterilized or at least 2 years postmenopausal) and who are not nursing may be included. Females who are childbearing potential may be included if they agree to avoid pregnancy during the study, and agree to use a birth control method.
9. Able to comply with schedule visits, treatment plan and study procedures.
10. Signed and dated informed consent indicating that the participant has been informed of all aspects of the study. In case of involuntary admission, a judge will consent the participant is capable to participate.

Exclusion Criteria:

1. History of suicide attempt in the previous year.
2. Not agree to abstain from cannabis.
3. Taking bupropion.
4. Recent (less than two months) myocardial infarction.
5. Previous adverse reaction that the investigator considers due to varenicline/nicotine patch and of sufficient concern that further exposure to varenicline/nicotine patch would be inadvisable.
6. Severe renal insufficiency.
7. Pregnancy or lactation.
8. Other severe acute or chronic medical or psychiatric condition that would make the subject inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of effectiveness: smoking abstinence rates | Between week 9 and week 16
  To compare smoking abstinence rates of varenicline relative to nicotine patch measured by CO-confirmed continuous abstinence rate.
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Randomization day
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 1
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 2
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 3
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 4
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 5
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 6
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 7
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 8
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 9
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 10
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 11
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 12
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Assessment of safety: incidence of emergent "severe" neuropsychiatric event | Week 13
  Differences in the incidence of emergent "severe" neuropsychiatric event. Solicited neuropsychiatric adverse events (AEs) will be collected by the use of Neuropsychiatric Adverse Event Interview (NAEI).
Psychiatric Evaluation done by a psychiatrist | From the screening day, on the randomization day, weekly during hospitalization (week 1 to week 4) and on the post-discharge weeks 5, 7, 9, 12 and 16.
  Psychiatric Evaluation done by a psychiatrist as a measure of Mental health assessment. Although psychiatric assessment will not use a specific tool, an interview with the patient will be delivered in order to assess psychopathology not covered by the instruments of the protocol, deepen in possible adverse events that may arise with the NAEI (Neuropsychiatric Adverse Event Interview) and readjust psychiatric medication if needed.
Clinical Global Impression of Severity (baseline) | It is assessed in the randomization day (day 1)
  The CGI-S is a clinician rated instrument measuring the severity of a subject's psychiatric condition on a 7 point scale at time of assessment, relative to clinician's past experience in patients with same diagnosis.
Clinical Global Impression of Improvement | During hospitalization, from week 1 to week 4, and on the post-discharge weeks 5, 7, 9, 12 and 16.
  The CGI-I is a clinician rated instrument that measures change in subject's psychiatric condition on a 7 point scale ranging from 1 (very much improved) to 7 (very much worse).
The Hospital Anxiety and Depression Scale (HADS) | From the randomization day, weekly during hospitalization (week 1 to week 4) and on the post-discharge weeks 5, 7, 9, 12 and 16.
  The Hospital Anxiety and Depression Scale (HADS) is a subject self-report scale and contains 14 items rated on 4-point Lickert-type scales. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression, being 0 not having anxiety or depression and 21 very anxious or depressed. The HADS uses a scale and therefore the data returned from the HADS is ordinal.
Columbia Suicide-Severity Rating Scale (C-SSRS) | From the screening day, on the randomization day, weekly during hospitalization (week 1 to week 4) and on the post-discharge weeks 5, 7, 9, 12 and 16.
  The Columbia Suicide-Severity Rating Scale (C-SSRS) rates an individual's degree of suicidal ideation which may be indicative of an individual's intent to complete suicide. It contains six "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past month and behaviors over their lifetime and past 3 months. Each question addresses a different component of the respondent's suicide ideation severity and behavior.
  1. wish to be dead
  2. non-specific suicidal thoughts 3-5: more specific suicidal thoughts and intent to act
  6: suicidal behavior over the respondent's lifetime and past 3 months
  An answer of "yes" to any of the six questions may indicate a need for referral to a trained mental health professional and an answer of "yes" to questions 4, 5 or 6 indicate high-risk.
Measurement of Nicotine Use Inventory (NUI) | From the randomization day, weekly during hospitalization (week 1 to week 4) and on the post-discharge weeks 5, 7, 9, 12, 14 and 16.
  The Measurement of Nicotine Use Inventory (NUI) is a questionnaire regarding use of cigarettes and other nicotine -containing products during the treatment period or tobacco products during the non-treatment period.
  The NUI consists of the following two questions: whether the person has smoked any cigarettes (even a puff) since the last contact and whether he has smoked any other tobacco products (eg, pipe, cigars, snuff, chew) since the last contact.
Minessota Nicotine Withdrawal Scale (MNWS) | From the randomization day, weekly during hospitalization (week 1 to week 4) and on the post-discharge weeks 5, 7, 9, 12 and 16.
  The Minessota Nicotine Withdrawal Scale (MNWS) is a subject self-report scale and contains 8 items (e.g., irritability, anxious, depressed mood, difficulty concentrating, increased appetite, insomnia, restless...) on a 5-point Lickert-type scales measuring nicotine withdrawal symptoms.
  Subjects were given a score on each item on a scale of 0 (not present) to 4 (severe). Summed (total) score excluding craving represent subject's symptoms of tobacco withdrawal, ranging from 0 to 32. We calculated a craving for tobacco score and a total score of withdrawal symptoms excluding craving. The higher score represent more sever craving and withdrawal.
Fagerström test for Cigarette Dependence (FTCD) | It is assessed in the randomization day (day 1)
  Cigarrette dependence was assessed using the Fagerström Test of Nicotine Dependence (FTND), which consists of six questions. Question 1 of the FTND read as follows: "How soon after you wake up do you smoke your first cigarette?" A total score was calculated as a sum of the six questions, with lower scores indicating lower dependence on nicotine: 0-2, very low dependence; 3-4, low dependence; 5, medium dependence; 6-7, high dependence; and 8-10, very high dependence.
End-expiratory exhaled carbon monoxid (exhaled CO) | From the randomization day, weekly during hospitalization (week 1 to week 4) and on the post-discharge weeks 5, 7, 9, 12 and 16.
  Breath carbon monoxide is the level of carbon monoxide in a person's exhalation. It can be measured in a breath carbon monoxide test, generally by using a carbon monoxide breath monitor (breath CO monitor), such as for motivation and education for smoking cessation and also as a clinical aid in assessing carbon monoxide poisoning.

CONTACTS AND LOCATIONS:
Overall Officials: Eugeni Bruguera, MD, Principal Investigator — Vall d'Hebron Institute of Research, Galatea Clinic; Dolores Braquehais, PhD, Principal Investigator — Galatea Clinic; Naia Sáez-Francàs, PhD, Principal Investigator — Sant Rafael Hospital; Cristina Pinet, MD, Principal Investigator — Hospital de Sant Pau; Gemma Nieva, PhD, Principal Investigator — Vall d'Hebron Institute of Research, Galatea Clinic
Locations (4):
- Spain (4):
  - Galatea Clinic, Barcelona
  - Sant Rafael Hospital, Barcelona
  - Vall d'Hebron Institute of Research, Barcelona
  - Hospital de Sant Pau, Barcelona

REFERENCES:
- [Background] Colton CW, Manderscheid RW. Congruencies in increased mortality rates, years of potential life lost, and causes of death among public mental health clients in eight states. Prev Chronic Dis. 2006 Apr;3(2):A42. Epub 2006 Mar 15. PMID 16539783
- [Background] Callaghan RC, Veldhuizen S, Jeysingh T, Orlan C, Graham C, Kakouris G, Remington G, Gatley J. Patterns of tobacco-related mortality among individuals diagnosed with schizophrenia, bipolar disorder, or depression. J Psychiatr Res. 2014 Jan;48(1):102-10. doi: 10.1016/j.jpsychires.2013.09.014. Epub 2013 Sep 27. PMID 24139811
- [Background] Prochaska JJ. Ten critical reasons for treating tobacco dependence in inpatient psychiatry. J Am Psychiatr Nurses Assoc. 2009 Dec;15(6):404-9. doi: 10.1177/1078390309355318. No abstract available. PMID 20336177
- [Background] Prochaska JJ, Fletcher L, Hall SE, Hall SM. Return to smoking following a smoke-free psychiatric hospitalization. Am J Addict. 2006 Jan-Feb;15(1):15-22. doi: 10.1080/10550490500419011. PMID 16449089
- [Background] Prochaska JJ, Hall SE, Delucchi K, Hall SM. Efficacy of initiating tobacco dependence treatment in inpatient psychiatry: a randomized controlled trial. Am J Public Health. 2014 Aug;104(8):1557-65. doi: 10.2105/AJPH.2013.301403. Epub 2013 Aug 15. PMID 23948001
- [Background] Hickman NJ, Prochaska JJ, Dunn LB. Screening for understanding of research in the inpatient psychiatry setting. J Empir Res Hum Res Ethics. 2011 Sep;6(3):65-72. doi: 10.1525/jer.2011.6.3.65. PMID 21931239
- [Background] Lasser K, Boyd JW, Woolhandler S, Himmelstein DU, McCormick D, Bor DH. Smoking and mental illness: A population-based prevalence study. JAMA. 2000 Nov 22-29;284(20):2606-10. doi: 10.1001/jama.284.20.2606. PMID 11086367
- [Background] Stockings EA, Bowman JA, Baker AL, Terry M, Clancy R, Wye PM, Knight J, Moore LH, Adams MF, Colyvas K, Wiggers JH. Impact of a postdischarge smoking cessation intervention for smokers admitted to an inpatient psychiatric facility: a randomized controlled trial. Nicotine Tob Res. 2014 Nov;16(11):1417-28. doi: 10.1093/ntr/ntu097. Epub 2014 Jun 17. PMID 24939916
- See also: Efficacy of a universal smoking cessation intervention initiated in inpatient psychiatry and continued post-discharge: A randomised controlled trial. — http://journals.sagepub.com/doi/10.1177/0004867417692424
- See also: Neuropsychiatric safety and efficacy of varenicline, bupropion, and nicotine patch in smokers with and without psychiatric disorders (EAGLES): a double-blind, randomised, placebo-controlled clinical trial. — http://dx.doi.org/10.1016/S0140-6736(16)30272-0